CLINICAL TRIAL: NCT05960955
Title: Phase II Clinical Study of Cadonilimab Combination With Chemotherapy With or Without the Anti-CD47 Antibody AK117 Neoadjuvant/Adjuvant Therapy for Resectable Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Cadonilimab Combination With Chemotherapy With or Without AK117 in Resectable Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK104-219
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Resectable Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Oxaliplatin; Docetaxel; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1 cohort 1 (Experimental): Subjects receive cadonilimab combination chemotherapy(SOX) neoadjuvant therapy 3 cycles.
  Interventions: Drug: Cadonilimab; Drug: Oxaliplatin; Drug: Tegafur-gimeracil-oteracil potassium
- Part 1 cohort 2 (Experimental): Subjects receive cadonilimab combination chemotherapy(SOX) and AK117 neoadjuvant therapy 3 cycles.
  Interventions: Drug: Cadonilimab; Drug: AK117; Drug: Oxaliplatin; Drug: Tegafur-gimeracil-oteracil potassium
- Part 2 cohort 1 (Experimental): Subjects receive cadonilimab combination chemotherapy(FLOT) neoadjuvant therapy 4 cycles.
  Interventions: Drug: Cadonilimab; Drug: Oxaliplatin; Drug: Docetaxel; Drug: 5-Fluorouracil
- Part 2 cohort 2 (Experimental): Subjects receive cadonilimab combination chemotherapy(FLOT) and AK117 neoadjuvant therapy 4 cycles.
  Interventions: Drug: Cadonilimab; Drug: AK117; Drug: Oxaliplatin; Drug: Docetaxel; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Cadonilimab — IV infusion,Specified dose on specified days
Drug: AK117 — IV infusion,Specified dose on specified days
  Arms: Part 1 cohort 2; Part 2 cohort 2
Drug: Oxaliplatin — IV infusion,Specified dose on specified days
Drug: Tegafur-gimeracil-oteracil potassium — Oral,Specified dose on specified days
  Arms: Part 1 cohort 1; Part 1 cohort 2
Drug: Docetaxel — IV infusion,Specified dose on specified days
  Arms: Part 2 cohort 1; Part 2 cohort 2
Drug: 5-Fluorouracil — IV infusion,Specified dose on specified days
  Arms: Part 2 cohort 1; Part 2 cohort 2

SUMMARY:
This trial is a Phase II study. All patients are resectable Gastric or Gastroesophageal Junction Adenocarcinoma, Eastern Cooperative Oncology Group (ECOG) performance status 0-1.The purpose of this study is to evaluate the efficacy and safety of cadonilimab combined with chemotherapy with or without AK117 neoadjuvantin treatment of resectable Gastric or Gastroesophageal Junction Adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide written informed consent.
* 18 to 75 years old.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has a histologically confirmed diagnosis of Gastric or Gastroesophageal Junction Adenocarcinoma(G/GEJ).
* Has Stage T3-4N+M0 G/GEJ (American Joint Committee on Cancer [AJCC])
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Has adequate organ function.

Exclusion Criteria:

* Are there suspected metastases or locally advanced, unresectable disease, regardless of disease stage.
* Is currently participating in a study of an investigational agent or using an investigational device.
* Has undergone major surgery within 30 days of Study Day 1.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* History of myocardial infarction, unstable angina, congestive heart failure within 12 months prior to day 1 of study treatment.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE), rate of surgical delays, abnormal laboratory findings of clinical significance | Up to approximately 2 years
Pathological complete response (pCR) rates | Up to approximately 2 years
  pCR is defined the 0% residual viable tumor cells in the primary tumor and sampled lymph nodes

SECONDARY OUTCOMES:
Major pathological response(MPR) rates | Up to approximately 2 years
  MPR is defined the ≤10% residual viable tumor cells in the primary tumor and sampled lymph nodes
Tumor regression grade(TRG) | Up to approximately 2 years
R0 resection rate | Up to approximately 2 years
Tumor descending stage rate | Up to approximately 2 years
  Proportion of subjects whose tumor TNM stage decreased from baseline before surgery
ORR | Up to approximately 2 years
EFS | Up to approximately 2 years
OS | Up to approximately 2 years
PK | Up to approximately 2 years
  Serum drug concentrations of cadonilimab and/or AK117 in individual subjects at different time points
ADA | Up to approximately 2 years
  Number of subjects with detectable anti-drug antibodies (ADA).

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Provincial Tumor Hospital, Tianjin, China